CLINICAL TRIAL: NCT03766048
Title: Non-inferiority Randomized Double Blind Controlled Trial Comparing Results of Laparoscopic Sacrocolpopexy With or Without Preventive Prerectal Mesh in Women Operated for Urogenital Prolapse Without Significant Posterior Vaginal Wall Prolapse
Brief Title: LAparoscopic Preventive PRErectal Mesh
Acronym: LAPREM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017_74; 2018-A01487-48 (Other: ID-RCB number, ANSM); PHRCN-17-0226 (Other: PHRC number, DGOS)
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Urogenital Prolapse
Keywords: Urogenital prolapse; laparoscopic sacropexy; mesh; medico-economic study
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-Anterior-Mesh, SAM (Experimental)
  Interventions: Procedure: Single-Anterior-Mesh, SAM
- Double-Mesh, DM (Sham Comparator)
  Interventions: Procedure: Double-Mesh, DM

INTERVENTIONS:
Procedure: Single-Anterior-Mesh, SAM — laparoscopic sacropexy is only performed with the anterior mes
  Arms: Single-Anterior-Mesh, SAM
Procedure: Double-Mesh, DM — laparoscopic sacropexy is performed using two synthetic non-absorbable meshes, both sutured to the promontory (Double-Mesh, DM): one mesh is placed in the vesicovaginal space and sutured to the uterine cervix or vaginal apex, and one mesh is placed in the rectovaginal space
  Arms: Double-Mesh, DM

SUMMARY:
Urogenital prolapse is a frequent and invalidating pathology in women, involving the anterior vaginal wall and the uterus in most cases. Posterior vaginal wall prolapse is present in only 50% of cases. Surgery is an option for women with troublesome prolapse. A woman's lifetime risk of undergoing surgery for pelvic organ prolapse (POP) surgery by the age of 80 is around 19%. Laparoscopic sacrocolpopexy (LS) with synthetic non-absorbable mesh is considered the gold standard, with a composite success rate of 85% at one year (Prospere study). Based on early experience and historical habits, a prerectal mesh was used to be systematically placed in the rectovaginal space, in addition to the anterior and apical mesh placed in the vesicovaginal space, in order to prevent de-novo posterior prolapse (reported rates up to 33%).

The benefit of preventive prerectal mesh is questionned on the basis of a single retrospective study comparing 68 LS with double-mesh (anterior & posterior, DM) to 32 LS with a single anterior mesh (SAM): posterior recurrence rates were respectively 5.9 vs. 31.3% (p<0,01), and total recurrence rates 16.2 vs. 43.8% (p<0.01). However, as this difference was not significant in the subgroup of patients without associated cervicocystopexy, the authors concluded that the risk of posterior failure was only due to the cervicocystopexy itself (anti-urinary incontinence procedure which has been abandoned since).

On the other hand, a prerectal mesh increases the risk for specific complications: rectal injury (up to 3%), anal pain (up to 25%), mesh exposition (up to 2%). Furthermore the posterior mesh increases the procedure by a minimum of 30 minutes (Robolaps study, unpublished data). The rate of de-novo obstructed defecation after LS with prerectal mesh is reported up to 25%. It could be explained by the mesh itself, but also by nerve injuries during the dissection of the rectovaginal space and rectal stalks.

ELIGIBILITY:
Inclusion Criteria:

* Women with a urogenital prolapse (anterior wall and/or uterus or vaginal apex) stage = 2 (Ba and/or C points ≥ - 1 cm using the POP-Q system),
* without significant posterior vaginal wall prolapse (Bp < -1 cm when apical prolapse is reduced using a retractor leaving the posterior vaginal wall free),

Exclusion Criteria:

* Previous surgical repair for Pelvic Organ Prolapse
* Any associated prolapse requiring any non-authorized additional surgical repair (Authorized additional surgical procedures are hysterectomy, ovariectomy, adnexectomy, salpingectomy, myomectomy, or suburethral vaginal tape.)
* Wish for future pregnancy
* Lack of health insurance
* Woman not reading French or unable to consent
* Woman under law protection

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with a urogenital prolapse for whom a laparoscopic sacrocolpopexy is planned.
Enrollment: 834 (Estimated)
Dates: Start 2019-09-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite criteria of success at 2 years follow-up | at 2 years after the intervention
  Composite criteria of success at 2 years follow-up: no symptom of vaginal bulge, no prolapse beyond the hymen (>0 cm), no reintervention for prolapse recurrence. Its advantage is that it considers only recurrences that are symptomatic or needing a reintervention. It is strongly linked with women satisfaction after prolapse surgery.

SECONDARY OUTCOMES:
Anatomical results | at 2 years
  Anatomical results will be based on clinical evaluation of patients at 2 years follow-up using the POP-Q system, with a specific evaluation of posterior vaginal wall with measures of the Bp point

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe LUCOT, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (9):
- France (9):
  - Hopital Estaing, Clermont-Ferrand
  - Ch Dunkerque, Dunkirk
  - Hopital Saint-Louis - La Rochelle, La Rochelle
  - Clinique Du Pre, Le Mans
  - Hop Jeanne de Flandre Chu Lille, Lille
  - Hopital Saint Vincent - Saint Antoine, Lille
  - Chu de Nice Hopital de L'Archet, Nice
  - Chu Nimes - Nimes, Nîmes
  - Chi Poissy St Germain Site de Poissy, Poissy